CLINICAL TRIAL: NCT05576012
Title: A Randomized, Double-Blind, Placebo-Controlled, First-in-Human Phase I Study Evaluating Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of SOL-116 in Healthy Subjects and Patients With Rheumatoid Arthritis
Brief Title: First in Human Study of a Monoclonal Antibody (SOL-116) Targeting BSSL (Bile Salt-Stimulated Lipase), Single and Multiple Dose Parts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lipum AB (Industry)
Collaborators: QPS Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPM-116-001
Record Dates: First submitted 2022-10-03; First posted 2022-10-12 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Part 1 single dose: Dose escalation in healthy subjects (up to 6 cohorts). Within each cohort, subjects will be randomized in a 3:1 ratio to receive either SOL-116 (n=6) or matching placebo (n=2) in a double-blind manner.
  Part 2 single dose in patients with rheumatoid arthritis (1 cohort). The patients will be randomized in a 3:1 ratio to receive either SOL-116 (n=6) or matching placebo (n=2) in a double-blind manner.
  Part 3 multiple dose in healthy subjects (1 or 2 cohorts). The subjects will be randomized in a 3:1 ratio to receive either SOL-116 (n=6) or matching placebo (n=2) in a double-blind manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOL-116 single dose (Parts 1 and 2); multiple dose (Part 3) (SC administration) (Experimental)
  Interventions: Biological: SOL-116
- Placebo single dose (Parts 1 and 2); multiple dose (Part 3) (SC administration) (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SOL-116 — Participants will receive SC injection in a double-blind manner
  Arms: SOL-116 single dose (Parts 1 and 2); multiple dose (Part 3) (SC administration)
Biological: Placebo — Participants will receive SC injection in a double-blind manner
  Arms: Placebo single dose (Parts 1 and 2); multiple dose (Part 3) (SC administration)

SUMMARY:
This is a randomized, double-blind, placebo-controlled, first-in-human phase I study. It consists of a single ascending dose part in healthy subjects (Part 1) and in patients with rheumatoid arthritis (Part 2) as well as a multiple dose part in healthy subjects (Part 3). The study will collect information on pharmacokinetics, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study and is willing and able to abide by the study restrictions.
2. Males and females aged between 18 and 65 years (inclusive) at Screening. For patients in the RA cohort, an age interval between 18 and 70 years (inclusive).
3. Normal clinically physical findings, apart from RA specific findings (including deviating laboratory values e.g., mild anaemia or swollen joints) for RA patients, including pulse rate, blood pressure, electrocardiogram (ECG), physical examination, and laboratory values (haematological/clinical chemistry) as judged by the Investigator. Healthy subjects must be negative for anti-CCP and have Rheumatoid Factor <1.5 ULN at Screening.
4. For Parts 1 and 3, body mass index (BMI) between 19.0 and 30.0 kg/m2 and body weight between 50 to 100 kg (inclusive) at Screening. For Part 2, body weight between 50 to 120 kg (inclusive) at Screening.
5. Sexually active male patients participating in the study must use a barrier method of contraception (condom) and refrain from sperm donation during the study and for at least 150 days after last dosing if their female sexual partner is of childbearing potential. Acceptable methods of birth control for female partners of male subjects are: hormonal contraceptives (oral contraceptives, implant or injection), intrauterine device (placed at least 1 month before the start of the study). Surgical sterilization of male patients can be accepted as a form of birth control if the sterilization procedure took place at least 6 months prior to the start of the study.
6. Females of childbearing potential must during the study and for at least 230 days after last dosing utilise a method of contraception that can achieve a failure rate of less than 1% per year when used consistently and correctly (defined in study protocol).
7. Females of non-childbearing potential must fulfil one of the following:

   * Irreversibly surgically sterile i.e., hysterectomy, bilateral salpingectomy, the fallopian tubes have been blocked or sealed (sterilization), and bilateral oophorectomy.
   * Spontaneous amenorrhoea during the last 12 months prior to enrolment, and having follicle stimulating hormone (FSH) levels in the postmenopausal range (i.e. ≥ 30 mIU/mL) at Screening.

   The following inclusion criterion is only applicable for RA patients:
8. Fulfilling the 2010 American College of Rheumatology (ACR)/European Union League Against Rheumatism (EULAR) classification criteria for RA [8].

   * Treatment with MTX for at least 12 weeks prior to treatment start and planned to continue with MTX during the study; if the MTX dose was changed during the 12-week period, such a patient may be included in the study based on Investigator judgement.
   * Patients naïve to biological disease modifying anti-rheumatic drug (bDMARD) or who are washed out (at least 5 half-lives) from such therapy before study drug dosing.
   * Patients naïve to conventional/targeted synthetic disease modifying anti-rheumatic drug (csDMARD/tsDMARD), except for MTX, or who are washed out since at least 12 weeks from such therapy before study drug dosing.
   * Use of oral glucocorticosteroids is allowed if equivalent to ≤5 mg/day of prednisolone on a stable dose for a least 4 weeks prior to dosing (Day 1) and expected to remain on that dose level for at least 4 weeks after dosing (Day 1).

Exclusion Criteria:

1. History of any clinically significant acute inflammatory joint disease (for the RA cohort; other than RA).
2. Any chronic or long-lasting disease which may interfere with the study objectives or jeopardise the safety of the subjects/patients as judged by the Investigator or responsible physician (for the RA cohort; other than RA).
3. Ongoing infection on Day-1.
4. Serious infection treated with antibiotics and evaluated by physician in the past 14 days prior to Day -1.
5. Current treatment with heparin products.
6. Use of any prescription or non-prescription drugs (excluding paracetamol, hormonal contraceptives), antacids, herbal, and dietary supplements (including St John's Wort) within 14 days (or 28 days if the drug is a potential hepatic enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug for healthy subjects and within 4 weeks prior to the first dose of study drug for RA patients, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject/patient safety. In RA patients, MTX and folic acid use are exempted.
7. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 2.0 times upper limit of normal (ULN); alkaline phosphatase and bilirubin ≥ 1.5 times the ULN at Screening or on Day -1. At screening, these assessments may be repeated once, at the discretion of the Investigator.
8. Serum creatinine > 1.5 times the ULN or eGFR <60 at Screening or on Day -1 (for Part 1 and Part 3). Estimated glomerular filtration rat (eGFR) <60 at Screening or on Day -1 (for Part 2). At Screening, these assessments may be repeated once, at the discretion of the Investigator.
9. Subjects/patients who have experienced surgery within 6 months of the screening visit that could negatively impact on the subject's/patient's participation in the opinion of a Principal Investigator or responsible physician.
10. High blood pressure at Screening or on Day -1, judged as clinically relevant by a Principal Investigator or responsible physician. A repeat test may be performed.
11. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV) at Screening.
12. Having evidence of active TB or latent TB at Screening as assessed by chest X-ray (RA patients only) and/or by QuantiFERON®-test. Applicable for RA patients only: in case of rescreening within three months after Screening, negative results from the initial chest X-ray and/or QuantiFERON®-test performed during Screening do not need to be repeated.
13. Subjects/patients who are currently enrolled in or have recently participated in another interventional clinical study defined as having received the last intervention within 90 days or 5 half-lives of the study drug (whichever is longer) prior to dosing (Parts 1 and 2) vs. prior to first dosing (Part 3) of the study drug.
14. History or known hypersensitivity or allergy, or any form of allergic reactions to any excipients in the study drug or to humanized or murine monoclonal antibodies (or immunoglobulins).
15. Receipt of a vaccine within 4 weeks (COVID-19 vaccine within 6 weeks) prior to dosing and/or the intention to receive a vaccine during the study. Deviation from this should be judged by the Investigator and in dialogue with the Sponsor.
16. Recent confirmed COVID-19 infection, with less than 6 weeks between recovery and dosing of study drug.
17. Blood or plasma donation within 3 months of enrolment.
18. Positive urine drug screen or alcohol test at Screening or on Day -1.
19. History of drug or alcohol abuse, at the discretion of the Investigator, within past 12 months prior to Screening.
20. The subject currently smokes or uses nicotine-containing products. Former smokers will be eligible, provided they have not smoked for at least 1 month prior to Screening. Positive cotinine test results at Screening or on Day -1 are reason for exclusion. Such positive test results can be repeated once to exclude environmental influence on the subject.
21. A positive pregnancy test or lactation at Screening or on Day -1.

    The following exclusion criteria are only applicable for RA patients:
22. Intra-articular or systemic corticosteroid injection within 4 weeks prior to dosing.
23. Current or expected need of other immunosuppressant medication except MTX and/or intra-articular corticosteroid injections.
24. Known Gilbert's syndrome or Screening laboratory values indicating Gilbert's syndrome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abd-Elaziz, MD, Principal Investigator — QPS Netherlands B.V.
Locations (2):
- Netherlands (2):
  - QPS Netherlands B.V., Groningen
  - CHDR (Stichting Centre for Human Drug Research), Leiden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a phase I study that covers three parts: ascending single doses in healthy subjects, single dose in patients and multiple doses in healthy subjects; each cohort is small 6 active + 2 placebo subjects. The complete results are found in the Clinical Study Report.
  In section Results Participant Flow, detailed design, dose levels, number of subjects are shown.
Groups:
- Cohort 1 (Active): 0.075 mg/kg SOL-116 (healthy subjects)
- Cohort 2 (Active): 0.225 mg/kg SOL-116 (healthy subjects)
- Cohort 3 (Active): 0.675 mg/kg SOL-116 (healthy subjects)
- Cohort 4 (Active): 2.025 mg/kg SOL-116 (healthy subjects)
- Cohort 5 (Active): 6.075 mg/kg SOL-116 (healthy subjects)
- Cohort 6 (Active): 3.0 mg/kg multiple dose (healthy subjects)
- Cohort 7 (Active): 2.025 mg/kg (patients with rheumatoid arthritis)
- Placebo (Cohort 1-5): Placebo (healthy subjects)
- Placebo (Cohort 6): Placebo, multiple dose (healthy subjects)
- Placebo (Cohort 7): Placebo (patients with rheumatoid arthritis)
Period: Overall Study
Arm/Group | Cohort 1 (Active) | Cohort 2 (Active) | Cohort 3 (Active) | Cohort 4 (Active) | Cohort 5 (Active) | Cohort 6 (Active) | Cohort 7 (Active) | Placebo (Cohort 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 (Single Dose): 0.075 mg/kg SOL-116 (healthy subjects)
- Cohort 2 (Single Dose): 0.225 mg/kg SOL-116 (healthy subjects)
- Cohort 3 (Single Dose): 0.675 mg/kg SOL-116 (healthy subjects)
- Cohort 4 (Single Dose): 2.025 mg/kg SOL-116 (healthy subjects)
- Cohort 5 (Single Dose): 6.075 mg/kg SOL-116 (healthy subjects)
- Cohort 6 (Multiple Doses): 3.0 mg/kg SOL-116 x 4 (healthy subjects)
- Cohort 7 (Single Dose): 2.025 mg/kg SOL-116 (patients with rheumatoid arthritis)
- Placebo (Coh 1-5): Placebo (Cohorts 1-5)
- Placebo (Cohort 6): Placebo (Cohorts 6)
- Placebo (Cohort 7): Placebo (Cohorts 7)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Coh 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (19.2) | 44.8 (17.1) | 42.8 (18.3) | 44.2 (14.4) | 45.5 (10.7) | 58.2 (3.7) | 58.2 (11.5) | 52.0 (14.3) | 57.5 (0.7) | 63.5 (0.7) | 50.0 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 2 | 4 | 4 | 3 | 3 | 0 | 1 | 23
  Male | 4 | 3 | 5 | 4 | 2 | 2 | 3 | 7 | 2 | 1 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 6 | 6 | 5 | 6 | 4 | 6 | 6 | 9 | 2 | 2 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  White | 5 | 6 | 5 | 5 | 5 | 5 | 5 | 7 | 1 | 2 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2 | 56

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability: Adverse Events
Description: Number of adverse events (AEs); (assessed as related and non-related)
Time Frame: From screening through study completion, day 90 (Cohorts 1-5 and 7) vs. day 169 (Cohort 6)
Population: Safety set
Measure: Number; unit: number of events
Groups:
- Cohort 3 (Single Dose): 0.675 mg/kg (healthy subjects)
- Placebo (Cohorts 1-5): Placebo (Cohorts 1-5)
- Placebo (Cohort 6): Placebo (Cohort 6)
- Placebo (Cohort 7): Placebo (Cohort 7), patients with rheumatoid arthritis
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Cohorts 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
number of events | 7 | 9 | 8 | 8 | 4 | 24 | 28 | 8 | 3 | 4

2. Primary Outcome: Safety and Tolerability: Injection Site Reactions
Description: Number of injection site reactions (dryness, redness, swelling, pain/tenderness and itching)
Time Frame: From screening through study completion, day 90 (Cohorts 1-5 and 7) vs. day 169 (Cohort 6)
Population: Safety set
Measure: Number; unit: number of events
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Cohorts 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
number of events | 0 | 0 | 1 | 4 | 3 | 0 | 3 | 2 | 0 | 0

3. Primary Outcome: Safety and Tolerability: Clinical Laboratory Evaluations
Description: Number of clinically significant laboratory abnormalities
Time Frame: From screening through study completion, day 90 (Cohorts 1-5 and 7) vs. day 169 (Cohort 6)
Population: Safety set
Measure: Count of Units; unit: samples
Units Other Than Participants: samples
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Cohorts 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
Number analyzed (samples) | 66 | 66 | 66 | 66 | 66 | 60 | 66 | 110 | 20 | 22
samples | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Safety and Tolerability: Immune Reactions
Description: Number of immune reactions (hypersensitivity, cytokine release syndrome, immunogenicity)
Time Frame: From screening through study completion, day 90 (Cohorts 1-5 and 7) vs. day 169 (Cohort 6)
Population: Safety set
Measure: Number; unit: events
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Cohorts 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Safety and Tolerability: Electrocardiogram (ECG)
Description: Number of clinically significant abnormal findings recorded by investigator based on HR, PR, QRS and QT values of ECG
Time Frame: From screening through study completion, day 90 (Cohorts 1-5 and 7) vs. day 169 (Cohort 6)
Population: Safety set
Measure: Number; unit: events
Units Other Than Participants: assessments
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Cohorts 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
Number analyzed (assessments) | 48 | 48 | 48 | 48 | 48 | 66 | 48 | 80 | 22 | 20
events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Safety and Tolerability: Vital Signs - Temporal Body Temperature
Description: Number of clinically significant abnormal findings - Temporal Body Temperature
Time Frame: From screening through study completion: screening, pre-dose, 1, 4, 24, 48, 72 hours and Days 14, 21, 49 and 90 (cohorts 1-5 and 7). For cohort 6: screening, pre-dose, 1, 4, 24, 72 hours and Days 8, 29, 57, 85, 86, 88, 92,169
Population: Safety set
Measure: Number; unit: events
Units Other Than Participants: assessments
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Coh 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
Number analyzed (assessments) | 66 | 66 | 66 | 66 | 66 | 84 | 66 | 110 | 28 | 22
events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Safety and Tolerability: Vital Signs - Pulse Rate
Description: Number of clinically significant abnormal findings - Pulse rate
Time Frame: as for outcome 6
Population: Safety set
Measure: Number; unit: events
Units Other Than Participants: assessments
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Coh 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
Number analyzed (assessments) | 66 | 66 | 66 | 66 | 66 | 84 | 66 | 110 | 28 | 22
events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Safety and Tolerability: Vital Signs - Blood Pressure
Description: Number of clinically significant abnormal findings - Blood pressure
Time Frame: as for outcome 6
Population: Safety set
Measure: Number; unit: events
Units Other Than Participants: assessments
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Coh 1-5) | Placebo (Cohort 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
Number analyzed (assessments) | 66 | 66 | 66 | 66 | 66 | 84 | 66 | 110 | 28 | 22
events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: PK Parameters for SOL-116: AUC0-inf
Description: Area under the concentration-time curve up to infinite time
Time Frame: Cohorts 1-5 and 7: Pre-dose, 1h, 4h, 8h, days 2, 3, 4, 8, 14, 21, 35, 49, 63 and 90. Cohort 6: Pre-dose, 4h, days 2, 4, 8, 11, 15, 29, 57, 85, 86, 88, 92, 95, 99, 113, 140, 154, 169
Population: Per-protocol set
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ug/mL | 418 (106) | 1110 (113) | 3930 (712) | 12300 (2380) | 30200 (6310) | 17500 (3810) | 11400 (5000)

10. Secondary Outcome: PK Parameters for SOL-116: AUC0-t
Description: Area under the concentration-time curve up to the last measurable concentration
Time Frame: as for outcome 9
Population: Per-protocol set
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ug/mL | 400 (105) | 1060 (121) | 3710 (641) | 11700 (2240) | 28900 (5600) | 8390 (1560) | 10100 (4710)

11. Secondary Outcome: PK Parameters for SOL-116: Cmax
Description: Maximal observed concentration (Cmax)
Time Frame: as for outcome 9
Population: Per-protocol set
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
ug/mL | 0.49 (0.18) | 1.28 (0.24) | 4.68 (1.08) | 16.30 (3.54) | 35.30 (11.10) | 34.60 (9.01) | 14.80 (3.36)

12. Secondary Outcome: PK Parameters for SOL-116: Tmax
Description: Time to Cmax
Time Frame: as for outcome 9
Population: Per-protocol set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 249 (129) | 220 (74) | 196 (59) | 122 (55) | 192 (49) | 159 (84) | 185 (85)

13. Secondary Outcome: PK Parameters for SOL-116: T1/2
Description: Outcome measure: Terminal elimination half-life
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 446 (41.8) | 459 (43.5) | 495 (62.7) | 465 (30.8) | 389 (110) | NA (NA) — Not estimated due to less than three measurable concentrations | 475 (106)

14. Secondary Outcome: PK Parameters for SOL-116: Vz/F
Description: Apparent volume of distribution following extravascular administration
Time Frame: as for outcome 9
Population: Per-protocol set
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
L | 9.58 (3.67) | 9.67 (2.83) | 10.20 (2.55) | 8.75 (2.21) | 7.59 (1.59) | NA (NA) — Not estimated due to less than three measurable concentrations | 11.50 (4.91)

15. Secondary Outcome: PK Parameters for SOL-116: CL/F
Description: Apparent total body clearance following extravascular administration
Time Frame: as for outcome 9
Population: Per-protocol set
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h | 0.0146 (0.0041) | 0.0145 (0.0029) | 0.0144 (0.0038) | 0.0130 (0.0031) | 0.0145 (0.0049) | 0.0125 (0.0021) | 0.0183 (0.0117)

16. Secondary Outcome: Immunogenicity Parameters: ADA
Description: Number of samples with detectable ADA (anti-drug antibodies)
Time Frame: Cohorts 1-5 and 7: Pre-dose, 4h, days 8, 21, 49 and 90. Cohort 6: Pre-dose, days 29, 57, 85, 113 and 169.
Population: Immunogenicity set
Measure: Number; unit: number of samples
Units Other Than Participants: samples
Groups:
- Placebo (Coh. 1-5): Placebo (Cohorts 1-5)
- Placebo (Coh. 6): Placebo (Cohort 6)
Arm/Group | Cohort 1 (Single Dose) | Cohort 2 (Single Dose) | Cohort 3 (Single Dose) | Cohort 4 (Single Dose) | Cohort 5 (Single Dose) | Cohort 6 (Multiple Doses) | Cohort 7 (Single Dose) | Placebo (Coh. 1-5) | Placebo (Coh. 6) | Placebo (Cohort 7)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 2
Number analyzed (samples) | 36 | 36 | 36 | 36 | 36 | 36 | 36 | 60 | 12 | 12
number of samples | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: In Parts 1 and 2 (single dose, Cohorts 1-5 and 7) follow-up was 90 days. In Part 3 (multiple doses, i.e., four doses, Cohort 6) follow-up was 169 days after first dose.
Groups:
- Cohort 1 (SOL-116); Cohort 2 (SOL-116); Cohort 3 (SOL-116); Cohort 4 (SOL-116); Cohort 5 (SOL-116); Cohorts 1-5 (Placebo): single dose
- Cohort 6 (SOL-116); Cohort 6 (Placebo): multiple doses
- Cohort 7 (SOL-116); Cohort 7 (Placebo): single dose, RA cohort
Arm/Group | Cohort 1 (SOL-116) | Cohort 2 (SOL-116) | Cohort 3 (SOL-116) | Cohort 4 (SOL-116) | Cohort 5 (SOL-116) | Cohort 6 (SOL-116) | Cohort 7 (SOL-116) | Cohorts 1-5 (Placebo) | Cohort 6 (Placebo) | Cohort 7 (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 3/6 | 5/6 | 3/6 | 5/6 | 6/6 | 6/10 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (SOL-116) (N=6) | Cohort 2 (SOL-116) (N=6) | Cohort 3 (SOL-116) (N=6) | Cohort 4 (SOL-116) (N=6) | Cohort 5 (SOL-116) (N=6) | Cohort 6 (SOL-116) (N=6) | Cohort 7 (SOL-116) (N=6) | Cohorts 1-5 (Placebo) (N=10) | Cohort 6 (Placebo) (N=2) | Cohort 7 (Placebo) (N=2)
Non st-segment elevation myocardial infarction (non-STEMI) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (SOL-116) (N=6) | Cohort 2 (SOL-116) (N=6) | Cohort 3 (SOL-116) (N=6) | Cohort 4 (SOL-116) (N=6) | Cohort 5 (SOL-116) (N=6) | Cohort 6 (SOL-116) (N=6) | Cohort 7 (SOL-116) (N=6) | Cohorts 1-5 (Placebo) (N=10) | Cohort 6 (Placebo) (N=2) | Cohort 7 (Placebo) (N=2)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (8) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Backpain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Backpain
Covid-19 (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Covid-19
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Dizziness
Flu (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cannula site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Swollen joints (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle tension (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter pylori infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flushes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT05576012/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT05576012/SAP_001.pdf